CLINICAL TRIAL: NCT06964906
Title: A Randomized, Open-Label, Blinded Endpoint Study of High-Intensity Focused Ultrasound (HIFU) Combined With Toripalimab Plus Chemotherapy Versus Chemotherapy as Neoadjuvant Therapy for Estrogen Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative (ER+/HER2-) Breast Cancer (NeoHunter)
Brief Title: Study of High-Intensity Focused Ultrasound (HIFU) Combined With Toripalimab Plus Chemotherapy Versus Chemotherapy as Neoadjuvant Therapy for Estrogen Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative (ER+/HER2-) Breast Cancer (NeoHunter)
Acronym: NeoHunter
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-0367
Record Dates: First submitted 2025-04-28; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: ER+/HER2- Breast Cancer
Keywords: Breast Neoplasms; High-intensity focused ultrasound; PD1; Toripalimab; nab-Paclitaxel; Epirubicin; Cyclophosphamide
MeSH Terms: conditions — Breast Neoplasms | interventions — toripalimab; 130-nm albumin-bound paclitaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIFU/Toripalimab + nab-P/Toripalimab + EC (Experimental): Participants receive HIFU treatment, followed by toripalimab (Q3W) + nab-Paclitaxel (QW) for 4 cycles (12 weeks), followed by toripalimab (Q3W) + epirubicin (Q3W) + cyclophosphamide (Q3W) for 4 cycles (12 weeks). Each cycle lasts 21 days.
  Interventions: Procedure: HIFU; Drug: Toripalimab; Drug: nab-Paclitaxel (nab-P); Drug: Epirubicin (E); Drug: Cyclophosphamide (C)
- nab-P/EC (Active Comparator): Participants receive nab-Paclitaxel (QW) for 4 cycles (12 weeks), followed by epirubicin (Q3W) + cyclophosphamide (Q3W) for 4 cycles (12 weeks). Each cycle lasts 21 days.
  Interventions: Drug: nab-Paclitaxel (nab-P); Drug: Epirubicin (E); Drug: Cyclophosphamide (C)

INTERVENTIONS:
Procedure: HIFU — HIFU therapy is administered to the targeted breast lesion site.
  Arms: HIFU/Toripalimab + nab-P/Toripalimab + EC
Drug: Toripalimab — 240 mg, IV infusion, Q3W
  Arms: HIFU/Toripalimab + nab-P/Toripalimab + EC
Drug: nab-Paclitaxel (nab-P) — 125 mg/m2, IV infusion, QW
Drug: Epirubicin (E) — 90 mg/m2, IV infusion, Q3W
Drug: Cyclophosphamide (C) — 600 mg/m2, IV infusion, Q3W

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of high-intensity focused ultrasound (HIFU) combined with toripalimab plus chemotherapy versus chemotherapy as neoadjuvant therapy for ER+/HER2- breast cancer.

DETAILED DESCRIPTION:
Study participants will be randomly allocated to either the experimental group or the control group and receive the following treatments. Experimental group: HIFU therapy followed by 8 cycles of neoadjuvant immunotherapy and chemotherapy; Control group: 8 cycles of neoadjuvant chemotherapy alone. Each cycle lasts 21 days. Subsequently, all participants will undergo surgery within 6 weeks after completion of neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 years.
2. Invasive breast cancer without distant metastasis, including either T1c-T2 (≥ 2 cm), cN1-cN2, or T3-T4, cN0-cN2.
3. Histopathologically confirmed ER-positive/HER2-negative, PR < 20% or Ki67 ≥ 20%, Grade 3 breast cancer.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Exclusion Criteria:

1. Female patients during pregnancy or lactation.
2. Diagnosis of bilateral breast cancer, occult breast cancer, or distant metastasis confirmed by pathology.
3. Has an active autoimmune disease that has received systemic treatment in the last 2 years.
4. Has a known history of human immunodeficiency virus (HIV), hepatitis B, or known active hepatitis C virus infection.
5. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
6. Has a known history of invasive malignancy that required systemic treatment in the last 5 years.
7. Uncontrolled concomitant diseases include severe infection, liver disease, cardiovascular disease, kidney disease, respiratory disease, diabetes, and others requiring systemic treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Pathological Complete Response (tpCR) Rate: ypT0/Tis, ypN0 | Up to approximately 30 weeks
  The tpCR rate is defined as the proportion of participants with no residual invasive cancer cells in both the breast primary tumor site (residual in situ cancer cells are permitted) and all sampled axillary lymph nodes.

SECONDARY OUTCOMES:
Breast Pathological Complete Response (bpCR) Rate: ypT0/Tis | Up to approximately 30 weeks
  The bpCR rate is defined as the proportion of participants with no residual invasive cancer cells in the breast primary tumor site (residual in situ cancer cells are permitted).
Objective Response Rate (ORR) | Up to approximately 30 weeks
  ORR is defined as the proportion of participants with a complete or partial response.
Event-Free Survival (EFS) | Approximately five years
  EFS is defined as the time from randomization to any of the following events: precludes surgery, local or distant recurrence, second primary malignancy, or death due to any cause.
Adverse Event (AE) | Approximately three years
  An AE is defined as any untoward medical occurrence in a study participant administered a medicinal product, temporally associated with study intervention, without presumption of causality.

CONTACTS AND LOCATIONS:
Overall Officials: Yiding Chen, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP